CLINICAL TRIAL: NCT04488367
Title: The Effects of the Timing of Tranexamic Acid Administration on Blood Loss in Hip Fractures.
Brief Title: Blood Loss After Early TXA in Hip Fractures.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Community Memorial Health System (Other)
Responsible Party: Principal Investigator, Michael Allen, Principal Investigator, Community Memorial Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TXARCT1
Record Dates: First submitted 2020-07-16; First posted 2020-07-28 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Hip Fractures
Keywords: tranexamic acid; TXA; hip fracture
MeSH Terms: conditions — Hip Fractures | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early TXA (Experimental): Experimental group will receive 10 mg/kg IV TXA while in the Emergency Department, and repeat preoperative and postoperative doses.
  Interventions: Drug: Tranexamic acid
- Control (Other): Control group will receive 100 mL 0.9% normal saline in the Emergency Department, and 10 mg/kg IV TXA before skin incision and again in post anesthesia care unit.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Tranexamic acid — 10 mg/kg IV TXA in the ED, repeat doses before skin incision and in PACU
  Other Names: Early TXA
  Arms: Early TXA
Drug: Normal Saline — 100 mL 0.9% normal saline in the ED, 10 mg/kg IV TXA before skin incision and in PACU
  Other Names: Control Placebo
  Arms: Control

SUMMARY:
Our present study aims to initiate TXA administration immediately upon diagnosis of hip fracture in the Emergency Department. This will be a single blind randomized controlled trial comparing early administration of TXA in the ED in addition to perioperative dosing versus the standard perioperative administration only. The study population will include patients who have sustained a femoral neck, intertrochanteric, or subtrochanteric femur fracture and are undergoing surgical internal fixation or arthroplasty. We will prospectively compare the need for blood transfusion, total and hidden blood loss, postoperative complications, length of stay and readmission within 30 days.

DETAILED DESCRIPTION:
Consent will be obtained for study enrollment from the patient or legal decision maker. The patient will then be randomized and stratified based on the fracture type, fixation method anticipated, and presence of anticoagulation.

Treatment drug and saline placebo will be blinded from the patient. Treatment arm patients will receive a dose of 10 mg/kg of TXA IV as soon as possible in the ED. They will then receive repeat doses prior to skin incision and again after the end of surgery. Control group will receive a placebo dose of normal saline in the ED and then the standard 10 mg/kg TXA doses prior to surgery and again after the end of surgery. The perioperative doses will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck, intertrochanteric, subtrochanteric femur fracture
* Age >18
* Undergoing surgical stabilization or arthroplasty by any method as determined by attending surgeon

Exclusion Criteria:

* Age <18
* Concomitant fracture
* Preoperative anemia needing blood transfusion before surgery
* Severe comorbidity (active cancer, severe pulmonary disease, ESRD)
* Allergy for tranexamic acid
* History of acute thromboembolic event (Deep Vein Thrombosis, Pulmonary Embolism, Stroke, TIA) in the previous 12 months
* Myocardial infarction in the previous 12 months
* Renal function impairment (creatinine clearance <30 mL/min), or kidney transplant
* History of hypercoagulability (Factor V Leiden, Protein C/S deficiency)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-07-06 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Change in calculated and recorded hemoglobin | From the time of randomization until discharge from the hospital after initial admission, or 4 weeks, whichever came first.
  Change in hemoglobin (blood loss) will be assessed based on preoperative blood draw and blood draws post op and on each inpatient day during hospitalization.
Total postoperative units of red blood cell transfusion | From the time of randomization until discharge from the hospital after initial admission, or 4 weeks, whichever came first.
  The number of units of RBC transfusions will be recorded and compared between treatment and placebo groups.

SECONDARY OUTCOMES:
VTE | Postoperative for 30 days
  DVT or PE
Infection | Postoperative for 30 days
  Superficial and deep infections
Readmission | Within 30 days postoperative
  30 day readmission
Other complications | Postoperative for 30 days
  Any additional unforeseen complications

CONTACTS AND LOCATIONS:
Overall Officials: Michael Allen, DO, Principal Investigator — Resident physician
Locations (1):
- Community Memorial Hospital, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foss NB, Kristensen MT, Kehlet H. Anaemia impedes functional mobility after hip fracture surgery. Age Ageing. 2008 Mar;37(2):173-8. doi: 10.1093/ageing/afm161. PMID 18349013
- [Background] Praetorius K, Madsen CM, Abrahamsen B, Jorgensen HL, Lauritzen JB, Laulund AS. Low Levels of Hemoglobin at Admission Are Associated With Increased 30-Day Mortality in Patients With Hip Fracture. Geriatr Orthop Surg Rehabil. 2016 Sep;7(3):115-20. doi: 10.1177/2151458516647989. Epub 2016 May 17. PMID 27551568
- [Background] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319
- [Background] Lei J, Zhang B, Cong Y, Zhuang Y, Wei X, Fu Y, Wei W, Wang P, Wen S, Huang H, Wang H, Han S, Liu S, Zhang K. Tranexamic acid reduces hidden blood loss in the treatment of intertrochanteric fractures with PFNA: a single-center randomized controlled trial. J Orthop Surg Res. 2017 Aug 15;12(1):124. doi: 10.1186/s13018-017-0625-9. PMID 28810918
- [Background] Baruah RK, Borah PJ, Haque R. Use of tranexamic acid in dynamic hip screw plate fixation for trochanteric fractures. J Orthop Surg (Hong Kong). 2016 Dec;24(3):379-382. doi: 10.1177/1602400322. PMID 28031511
- [Background] Baskaran D, Rahman S, Salmasi Y, Froghi S, Berber O, George M. Effect of tranexamic acid use on blood loss and thromboembolic risk in hip fracture surgery: systematic review and meta-analysis. Hip Int. 2018 Jan;28(1):3-10. doi: 10.5301/hipint.5000556. PMID 28983887
- [Background] Tian S, Shen Z, Liu Y, Zhang Y, Peng A. The effect of tranexamic acid on hidden bleeding in older intertrochanteric fracture patients treated with PFNA. Injury. 2018 Mar;49(3):680-684. doi: 10.1016/j.injury.2018.01.026. Epub 2018 Feb 2. PMID 29426608